CLINICAL TRIAL: NCT04336657
Title: COVID-19-Like Illness: Did we Have Unusual Severe Respiratory Tract Infections October-December 2019 Before WHO Announcement ?
Brief Title: Corona-Like Illness: Did we Got it Before WHO Announcement of the Disease?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU11
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: COVID-19; Corona-like illness; WHO announcement; Survey; IgG
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Survey to identify number of people who got unusual severe flu- like illness in last October- November
Diagnostic Test: IgG — Measure the past immunity of the disease (if possible)

SUMMARY:
A pneumonia of unknown cause detected in Wuhan, China was first reported to the WHO Country Office in China on 31 December 2019. The outbreak was declared a Public Health Emergency of International Concern on 30 January 2020. The spread and severity of the disease is variable from one country to another. Our team as well as many reports suggested that in some countries a " Flu like illness but much worse" was described in October, November and early in December before the WHO announcement. Was it COVID-19?

ELIGIBILITY:
Inclusion Criteria:

* All subject except excluded group

Exclusion Criteria:

* subject diagnosed as COVID-19 positive and their contacts

Ages: 8 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The survey will be distributed online in English and Arabic and all responders well be included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Measure frequency of people suffered from unusual flu-like symptoms before December 2019 | one month
  fever, dry cough, dyspnea, malaise, headache

SECONDARY OUTCOMES:
Measure remote immunity for COVID-19 in subject with past history of severe flu before WHO announcement date- if possible | 3 month
  serum IgG

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided